CLINICAL TRIAL: NCT04482062
Title: Edwards EVOQUE Transcatheter Tricuspid Valve Replacement: Pivotal Clinical Investigation of Safety and Clinical Efficacy Using a Novel Device
Brief Title: TRISCEND II Pivotal Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-05
Record Dates: First submitted 2020-07-09; First posted 2020-07-22 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Tricuspid Valve Regurgitation; Tricuspid Valve Insufficiency; Tricuspid Valve Disease; Heart Valve Diseases; Cardiovascular Diseases; Heart Failure
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases; Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Edwards EVOQUE System & OMT (Experimental): Transcatheter tricuspid valve replacement with the Edwards EVOQUE System in conjunction with optimal medical therapy (OMT) in patients with tricuspid regurgitation
  Interventions: Device: Edwards EVOQUE System
- Optimal Medical Therapy (OMT) (Active Comparator): Optimal medical therapy (OMT) alone in patients with tricuspid regurgitation
  Interventions: Drug: Optimal Medical Therapy
- Single-Arm Registry (Experimental): Transcatheter tricuspid valve replacement with the Edwards EVOQUE System in conjunction with optimal medical therapy (OMT) in patients with tricuspid regurgitation who are not eligible for randomization
  Interventions: Device: Edwards EVOQUE System
- Continued Access Study (Experimental): Provides continued access to transcatheter tricuspid valve replacement with the Edwards EVOQUE System in conjunction with optimal medical therapy (OMT) in patients with tricuspid regurgitation.
  Interventions: Device: Edwards EVOQUE System

INTERVENTIONS:
Device: Edwards EVOQUE System — Transcatheter tricuspid valve replacement with the Edwards EVOQUE System in conjunction with OMT
  Other Names: Transcatheter tricuspid valve replacement
  Arms: Continued Access Study; Edwards EVOQUE System & OMT; Single-Arm Registry
Drug: Optimal Medical Therapy — Optimal Medical Therapy
  Arms: Optimal Medical Therapy (OMT)

SUMMARY:
Pivotal trial to evaluate the safety and effectiveness of the Edwards EVOQUE tricuspid valve replacement system

DETAILED DESCRIPTION:
The study is a prospective, multi-center, randomized controlled pivotal clinical trial to evaluate the safety and effectiveness of the EVOQUE System with optimal medical therapy (OMT) compared to OMT alone in the treatment of patients with at least severe tricuspid regurgitation. Subjects will be followed at discharge, 30 days, 3 months, 6 months and annually through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Despite medical therapy (OMT) per the local Heart Team, patient has signs of TR, symptoms from TR, or prior heart failure hospitalization from TR. Patient must be on OMT per the local heart team at the time of TR assessment for trial eligibility (TTE). OMT includes stable oral diuretic medications, unless patient has a documented history of intolerance.
* Functional and/or degenerative TR graded as at least severe on a transthoracic echocardiogram (assessed by the echo core lab using a 5-grade classification)
* The Local Heart Team determines that the patient is appropriate for transcatheter tricuspid valve replacement
* Patient is willing and able to comply with all study evaluations and provides written informed consent.

Exclusion Criteria:

* Anatomy precluding proper device delivery, deployment and/or function
* LVEF < 25%
* Evidence of severe right ventricular dysfunction
* Any of the following pulmonary pressure parameters:

  1. PASP >60 mmHg by echo Doppler (unless RHC demonstrates PASP ≤70 mmHg)
  2. PASP >70 mmHg by RHC
  3. PVR >5 Wood units by RHC (unless PVR ≤5 Wood units and systolic BP >85 mmHg after vasodilator challenge)
* Previous tricuspid surgery or intervention
* Presence of trans-tricuspid pacemaker or defibrillator lead with any of the following:

  1. Implanted in the RV within the last90 days
  2. Patient is pacemaker dependent5 on trans-tricuspid lead without alternative pacing option
  3. Has delivered appropriate ICD therapy
* Severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation.
* Active endocarditis within the last 90 days or infection requiring antibiotic therapy (oral or intravenous) within the last 14 days
* Hemodynamically significant pericardial effusion
* Significant intra-cardiac mass, thrombus, or vegetation.
* Clinically significant, untreated coronary artery disease requiring revascularization, evidence of acute coronary syndrome, recent myocardial infarction within the last 30 days.
* Any of the following cardiovascular procedures:

  1. Percutaneous coronary, intracardiac, or endovascular intervention within the last 30 days
  2. Carotid surgery within the last 30 days
  3. Direct current cardioversion within the last 30 days
  4. Leadless RV pacemaker implant within the last 30 days
  5. Cardiac surgery within the last 90 days
* Known history of untreated severe symptomatic carotid stenosis (>50% by ultrasound) or asymptomatic carotid stenosis (>70% by ultrasound)
* Need for emergent or urgent surgery for any reason, any planned cardiac surgery within the next 12 months (365days), or any planned percutaneous cardiac procedure within the next 90 days
* Hypotension (systolic pressure <90 mmHg) or requirement for inotropic support or hemodynamic support within the last 30 days
* Patient with refractory heart failure requiring or which required advanced intervention (i.e. left ventricular assist device, transplantation) (ACC/AHA/ESC/EACTS Stage D heart failure)
* Deep vein thrombosis (DVT) or pulmonary embolism (PE) in the last 6 months (180 days)
* Stroke within the last 90 days
* Modified Rankin Scale ≥ 4 disability
* Severe renal insufficiency with estimated glomerular filtration rate (eGFR) ≤ 25 mL/min/1.73m2 or requiring chronic renal replacement therapy.
* Patients with hepatic insufficiency or cirrhosis with Child-Pugh score class C
* Patient is oxygen-dependent or requires continuous home oxygen
* Chronic anemia with transfusion dependency or Hgb < 9 g/dL not corrected by transfusion
* Unable to walk at least 100 meters in a 6-minute walk test
* Thrombocytopenia (Platelet count < 75,000/mm3) or thrombocytosis (Platelet count > 750,000/mm3)
* Known bleeding or clotting disorders or patient refuses blood transfusion
* Active gastrointestinal (GI) bleeding within the last 90 days
* Pregnant, breastfeeding, or planning pregnancy within the next 12 months (365 days).
* Patients in whom (any of the following):

  1. TEE is contraindicated or cannot be completed
  2. tricuspid valve anatomy is not evaluable by TTE or TEE
* In the opinion of the investigator, access to and through the femoral vein/IVC with a guide sheath and delivery catheter is deemed not feasible (e.g. occluded femoral veins, occluded or thrombosed IVC filter)
* Untreatable hypersensitivity or contraindication to any of the following: all antiplatelets, all anticoagulants, nitinol alloys (nickel and titanium), bovine tissue, glutaraldehyde, or contrast media
* Currently participating in another investigational biologic, drug or device study
* Co-morbid condition(s) that, in the opinion of the Investigator, limit life expectancy to < 12 months (365 days).
* Presence of infiltrative cardiomyopathy or valvulopathy (including carcinoid, amyloidosis, sarcoidosis, hemochromatosis) or significant uncorrected congenital heart disease (including but not limited to hemodynamically significant atrial septal defect, RV dysplasia, and arrhythmogenic RV)
* Any condition, in the opinion of the investigator, making it unlikely the patient will be able to complete all protocol procedures and follow-ups
* Other medical, social, or psychological conditions that preclude appropriate consent and follow-up, including patients under guardianship
* Any patient considered to be vulnerable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1070 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2030-06-27 (Estimated)

PRIMARY OUTCOMES:
Randomized Cohort: Tricuspid Regurgitation (TR) grade reduction | 6 months
  Comparison of number of participants with reduction in TR between experimental and active comparator arms. TR severity will be assessed using the 5-grade scale with the addition of "none/trace" to represent the lack of TR (scale: none/trace, mild, moderate, severe, massive, torrential). Lower grades of TR are better.
Randomized Cohort: Hierarchical composite endpoint including: Kansas City Cardiomyopathy Questionnaire (KCCQ) improvement, New York Heart Association (NYHA) functional class improvement, and 6-minute walk test distance improvement | 6 months
  Comparison of number of wins with composite endpoint event improvement between experimental and active comparator arms
Randomized Cohort: Rate of Major Adverse Events (MAE) | 30 days
  Rate of Major Adverse Events (MAE) in experimental arm (Edwards EVOQUE System & OMT)
Randomized Cohort: Hierarchical composite endpoint: all-cause mortality, RVAD implantation or heart transplant, tricuspid valve intervention, heart failure hospitalizations, KCCQ improvement, NYHA functional class improvement, and 6MWD improvement | 1 year
  Comparison of number of wins with composite endpoint events or improvement between experimental and active comparator arms
Continued Access Study: Rate of Major Adverse Events (MAE) | 30 days
  Rate of MAEs in the Continued Access Study arm
Continued Access Study: Tricuspid Regurgitation (TR) grade reduction to moderate, mild, or none/trace | 6 months
  TR grade reduction to moderate, mild, or none/trace from baseline. TR severity will be assessed using the 5-grade scale with the addition of "none/trace" to represent the lack of TR (scale: none/trace, mild, moderate, severe, massive, torrential); Lower grades of TR are better.
Continued Access Study: Quality of Life (QOL) as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 6 months
  Improvement in QOL (by KCCQ overall summary score) of at least 10 points. KCCQ overall summary score is a patient-reported measure of health status, ranging from 0 to 100, where higher scores reflect better QOL.
Continued Access Study: New York Heart Association (NYHA) functional class | 6 months
  NYHA functional class improvement of at least 1 class. NYHA functional classification system categorizes heart failure patients into 4 classes based on physical activity limitation and symptom severity: class I (no symptoms and no limitation in ordinary physical activity), class II (mild symptoms and slight limitation during ordinary activity), class III (marked limitation in activity due to symptoms, even during less-than-ordinary activity; comfortable only at rest, and class IV (severe limitations; experiences symptoms even while at rest).
Continued Access Study: 6MWD | 6 months
  6MWD improvement of at least 30 meters
Continued Access Study: All-cause mortality | 1 year
  Deaths from any cause
Continued Access Study: Durable right ventricular assist device (RVAD) implantation or heart transplant | 1 year
  Durable RVAD implantation or heart transplant
Continued Access Study: Total number of patients requiring tricuspid valve surgery or percutaneous tricuspid intervention | 1 year
  Total number of patients requiring tricuspid valve surgery or percutaneous tricuspid intervention.
Continued Access Study: Annualized rate of heart failure hospitalizations | 1 year
  Annualized rate of heart failure hospitalizations
Continued Access Study: Quality of Life (QOL) as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 1 year
  Improvement in QOL (by KCCQ overall summary score) of at least 10 points. KCCQ overall summary score is a patient-reported measure of health status, ranging from 0 to 100, where higher scores reflect better QOL.
Continued Access Study: New York Heart Association (NYHA) functional class | 1 year
  NYHA functional class improvement of at least 1 class. NYHA functional classification system categorizes heart failure patients into 4 classes based on physical activity limitation and symptom severity: class I (no symptoms and no limitation in ordinary physical activity), class II (mild symptoms and slight limitation during ordinary activity), class III (marked limitation in activity due to symptoms, even during less-than-ordinary activity; comfortable only at rest, and class IV (severe limitations; experiences symptoms even while at rest).
Continued Access Study: 6MWD | 1 year
  6MWD improvement of at least 30 meters

SECONDARY OUTCOMES:
Randomized cohort: Tricuspid Regurgitation (TR) grade reduction | Time Frame: Discharge (assessed up to 7 days post procedure)
  TR grade reduction from baseline to discharge (assessed up to 7 days post procedure). TR severity will be assessed using the 5-grade scale with the addition of "none/trace" to represent the lack of TR (scale: none/trace, mild, moderate, severe, massive, torrential). Lower grades of TR are better.
Randomized cohort: All-Cause Mortality | 1 year, annually through 5 years
  Total number of deaths from any cause
Randomized cohort: Heart failure hospitalizations | 1 year, annually through 5 years
  Total number of patients with at least one hospital admission due to heart failure
Randomized cohort: Non-elective tricuspid valve re-intervention (percutaneous or surgical) | 1 year, annually through 5 years
  Total number of patients with at least one non-elective tricuspid valve re-intervention
Randomized cohort: Durable RVAD implantation or heart transplant | 1 year, annually through 5 years
  Total number of patients requiring RVAD implantation or heart transplant
Randomized cohort: Need for paracentesis | 1 year, annually through 5 years
  Total number of patients who required paracentesis
Randomized cohort: Reduction in TR grade by at least one grade | 1 year
  Total number of patients with at least one grade TR reduction
Randomized cohort: Reduction in New York Heart Association (NYHA) functional class by at least one grade | 1 year
  Total number of patients with NYHA functional class improvement of at least 1 class. The NYHA functional classification system categorizes heart failure patients into 4 classes based on physical activity limitation and symptom severity: class I (no symptoms and no limitation in ordinary physical activity), class II (mild symptoms and slight limitation during ordinary activity), class III (marked limitation in activity due to symptoms, even during less-than-ordinary activity; comfortable only at rest, and class IV (severe limitations; experiences symptoms even while at rest).
Randomized cohort: Change in Quality of Life (QOL) as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline | 1 year
  Change in QOL (by KCCQ overall summary score) of at least 10 points. KCCQ overall summary score is a patient-reported measure of health status, ranging from 0 to 100, where higher scores reflect better QOL.
Randomized cohort: Death and heart failure hospitalization | 1 year
  Comparison of number of wins with death and HFH between experimental and active comparator arms
Randomized cohort: All-cause hospitalizations | 1 year
  Total number of patients with hospitalizations from any cause
Randomized cohort: All-cause mortality | 1 year
  Total number of patients with deaths from any cause
Randomized cohort: Change in 6MWD from baseline | 1 year
  Change in 6MWD from baseline
Roll-in cohort: Tricuspid Regurgitation (TR) grade reduction | Time Frame: Discharge (assessed up to 7 days post procedure)
  TR grade reduction from baseline to discharge (assessed up to 7 days post procedure). TR severity will be assessed using the 5-grade scale with the addition of "none/trace" to represent the lack of TR (scale: none/trace, mild, moderate, severe, massive, torrential). Lower grades of TR are better.
Roll-in cohort: All-cause mortality | 1 year, annually through 5 years
  Total number of deaths from any cause
Roll-in cohort: Heart failure hospitalizations | 1 year, annually through 5 years
  Total number of hospital admissions due to heart failure
Roll-in cohort: Non-elective tricuspid valve re-intervention (percutaneous or surgical) | 1 year, annually through 5 years
  Total number of non-elective tricuspid valve re-interventions
Roll-in cohort: Durable RVAD implantation or heart transplant | 1 year, annually through 5 years
  Total number of patients requiring RVAD implantation or heart transplant
Roll-in cohort: Need for paracentesis | 1 year, annually through 5 years
  Total number of patients who required paracentesis
Roll-in cohort: Reduction in tricuspid regurgitation (TR) grade by at least one grade | 1 year
  Total number of patients with at least one grade TR reduction. TR severity will be assessed using the 5-grade scale with the addition of "none/trace" to represent the lack of TR (scale: none/trace, mild, moderate, severe, massive, torrential). Lower grades of TR are better.
Roll-in cohort: Reduction in New York Heart Association (NYHA) functional class by at least one grade | 1 year
  Total number of patients with NYHA functional class improvement of at least 1 class. The NYHA functional classification system categorizes heart failure patients into 4 classes based on physical activity limitation and symptom severity: class I (no symptoms and no limitation in ordinary physical activity), class II (mild symptoms and slight limitation during ordinary activity), class III (marked limitation in activity due to symptoms, even during less-than-ordinary activity; comfortable only at rest, and class IV (severe limitations; experiences symptoms even while at rest).
Roll-in cohort: Change in Quality of Life (QOL) as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline | 1 year
  Change in QOL (by KCCQ overall summary score) of at least 10 points. KCCQ overall summary score is a patient-reported measure of health status, ranging from 0 to 100, where higher scores reflect better QOL.
Roll-in cohort: Death and heart failure hospitalization | 1 year
  Total number of patients with death or heart failure hospitalization
Roll-in cohort: All-cause hospitalizations | 1 year
  Total number of patients with hospitalizations from any cause
Roll-in cohort: All-cause mortality | 1 year
  Total number of patients with deaths from any cause
Roll-in cohort: Change in 6MWD from baseline | 1 year
  Change in 6MWD from baseline
Registry cohort: Tricuspid Regurgitation (TR) grade reduction | Time Frame: Discharge (assessed up to 7 days post procedure)
  TR grade reduction from baseline to discharge. TR severity will be assessed using the 5-grade scale with the addition of "none/trace" to represent the lack of TR (scale: none/trace, mild, moderate, severe, massive, torrential). Lower grades of TR are better.
Registry cohort: All-cause mortality | 1 year, annually through 5 years
  Total number of deaths from any cause
Registry cohort: Heart failure hospitalizations | 1 year, annually through 5 years
  Total number of hospital admissions due to heart failure
Registry cohort: Change in 6MWD from baseline | 1 year
  Change in 6MWD from baseline
Registry cohort: Non-elective tricuspid valve re-intervention (percutaneous or surgical) | 1 year, annually through 5 years
  Total number of non-elective tricuspid valve re-interventions
Registry cohort: Durable RVAD implantation or heart transplant | 1 year, annually through 5 years
  Total number of patients requiring RVAD implantation or heart transplant
Registry cohort: Need for paracentesis | 1 year, annually through 5 years
  Total number of patients who required paracentesis
Registry cohort: Reduction in TR grade by at least one grade | 1 year
  Total number of patients with at least one grade TR reduction
Registry cohort: Reduction in New York Heart Association (NYHA) functional class by at least one grade | 1 year
  Total number of patients with NYHA functional class improvement of at least 1 class. The NYHA functional classification system categorizes heart failure patients into 4 classes based on physical activity limitation and symptom severity: class I (no symptoms and no limitation in ordinary physical activity), class II (mild symptoms and slight limitation during ordinary activity), class III (marked limitation in activity due to symptoms, even during less-than-ordinary activity; comfortable only at rest, and class IV (severe limitations; experiences symptoms even while at rest).
Registry cohort: Change in Quality of Life (QOL) as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline | 1 year
  Change in QOL (by KCCQ overall summary score) of at least 10 points. KCCQ overall summary score is a patient-reported measure of health status, ranging from 0 to 100, where higher scores reflect better QOL.
Registry cohort: Death and heart failure hospitalization | 1 year
  Total number of patients with death and heart failure hospitalization
Registry cohort: All-cause hospitalizations | 1 year
  Total number of patients with hospitalizations from any cause
Registry cohort: All-cause mortality | 1 year
  Total number of patients with deaths from any cause
Continued Access Study: Tricuspid Regurgitation (TR) grade reduction | Time Frame: Discharge (assessed up to 7 days post procedure)
  TR grade reduction from baseline to discharge. TR severity will be assessed using the 5-grade scale with the addition of "none/trace" to represent the lack of TR (scale: none/trace, mild, moderate, severe, massive, torrential). Lower grades of TR are better.
Continued Access Study: All-cause mortality | 1 year, annually through 5 years
  Total number of deaths from any cause
Continued Access Study: Heart failure hospitalizations | 1 year, annually through 5 years
  Total number of hospital admissions due to heart failure
Continued Access Study: Non-elective tricuspid valve re-intervention (percutaneous or surgical) | 1 year, annually through 5 years
  Total number of non-elective tricuspid valve re-interventions
Continued Access Study: Durable RVAD implantation or heart transplant | 1 year, annually through 5 years
  Total number of patients requiring RVAD implantation or heart transplant
Continued Access Study: Need for paracentesis | 1 year, annually through 5 years
  Total number of patients who required paracentesis

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hahn, MD, Principal Investigator — Columbia University; Susheel Kodali, MD, Principal Investigator — Columbia University; Philipp Lurz, MD, Principal Investigator — Herzzentrum Leipzig GmbH; Vinod Thourani, MD, Principal Investigator — Piedmont Heart Institute
Locations (62):
- United States (55):
  - SJHMC Heart and Vascular Institute, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Florida Heart & Vascular Care - JFK, Atlantis, Florida
  - The Cardiac & Vascular Institute Research Foundation, Gainesville, Florida
  - NCH Heart Institute, Naples, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Ascension Via Christi St. Francis, Wichita, Kansas
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Hospital and Health Systems, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - State University of New York at Buffalo, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medicine-New York Presbyterian Hospital, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lankenau Heart Institute, Wynnewood, Pennsylvania
  - Saint Thomas Health, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - HCA Houston Healthcare, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor Heart Hopsital Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Mason Franciscan Health, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
- Germany (7):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen, Bad Oeynhausen
  - Herzzentrum Universitätsklinik Bonn, Bonn
  - Herzzentrum der Uniklinik Köln, Cologne
  - Herzzentrum Dresden Universitätsklinik, Dresden
  - Herzzentrum Leipzig GmbH, Leipzig
  - Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität München - Großhadern, München

REFERENCES:
- [Derived] Arnold SV, Hahn RT, Thourani VH, Makkar R, Makar M, Sharma RP, Haeffele C, Davidson CJ, Narang A, O'Neill B, Lee J, Yadav P, Zahr F, Chadderdon S, Eleid M, Pislaru S, Smith R, Szerlip M, Whisenant B, Sekaran N, Garcia S, Stewart-Dehner T, Grayburn PA, Sannino A, Snyder C, Zhang Y, Mack MJ, Leon MB, Lurz P, Kodali S, Cohen DJ; TRISCEND II Pivotal Trial Investigators. Quality of Life After Transcatheter Tricuspid Valve Replacement: 1-Year Results From TRISCEND II Pivotal Trial. J Am Coll Cardiol. 2025 Jan 28;85(3):206-216. doi: 10.1016/j.jacc.2024.10.067. Epub 2024 Oct 30. PMID 39480380
- [Derived] Hahn RT, Makkar R, Thourani VH, Makar M, Sharma RP, Haeffele C, Davidson CJ, Narang A, O'Neill B, Lee J, Yadav P, Zahr F, Chadderdon S, Eleid M, Pislaru S, Smith R, Szerlip M, Whisenant B, Sekaran NK, Garcia S, Stewart-Dehner T, Thiele H, Kipperman R, Koulogiannis K, Lim DS, Fowler D, Kapadia S, Harb SC, Grayburn PA, Sannino A, Mack MJ, Leon MB, Lurz P, Kodali SK; TRISCEND II Trial Investigators. Transcatheter Valve Replacement in Severe Tricuspid Regurgitation. N Engl J Med. 2025 Jan 9;392(2):115-126. doi: 10.1056/NEJMoa2401918. Epub 2024 Oct 30. PMID 39475399
- [Derived] Kodali S, Hahn RT, George I, Davidson CJ, Narang A, Zahr F, Chadderdon S, Smith R, Grayburn PA, O'Neill WW, Wang DD, Herrmann H, Silvestry F, Elmariah S, Inglessis I, Passeri J, Lim DS, Salerno M, Makar M, Mack MJ, Leon MB, Makkar R; TRISCEND Investigators. Transfemoral Tricuspid Valve Replacement in Patients With Tricuspid Regurgitation: TRISCEND Study 30-Day Results. JACC Cardiovasc Interv. 2022 Mar 14;15(5):471-480. doi: 10.1016/j.jcin.2022.01.016. PMID 35272771
- [Derived] Lurz P, Kresoja KP. Tricuspid Valve Therapies: Closing the Gap. JACC Cardiovasc Interv. 2021 Jun 14;14(11):1241-1242. doi: 10.1016/j.jcin.2021.04.008. No abstract available. PMID 34112461